CLINICAL TRIAL: NCT01815307
Title: Randomized Phase II Study of Gemcitabine Versus S-1 Adjuvant Therapy After Hemihepatectomy for Biliary Tract Cancer
Brief Title: Phase II Study of Gemcitabine Versus S-1 Adjuvant Therapy After Hemihepatectomy for Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHBO1208; UMIN000009945 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-03-05; First posted 2013-03-21 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2017-09

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine group (Experimental): 1000mg/m2, day 1 every 2 weeks
  Interventions: Drug: Gemcitabine
- S-1 group (Experimental): 80mg/m2/day, day 1-28, every 6 weeks
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2, day 1 every 2 weeks
  Other Names: gemzer
  Arms: Gemcitabine group
Drug: S-1 — 80mg/m2/day, day 1-28, every 6 weeks
  Other Names: TS-1
  Arms: S-1 group

SUMMARY:
To compare efficacy and safety of Gemcitabine versus S-1 adjuvant therapy after hemihepatectomy.

DETAILED DESCRIPTION:
There is no standard adjuvant therapy after liver hemi-hepatectomy due to bile duct cancer, because of high surgical morbidity ratio and high adverse event ratio of adjuvant therapy. For example, our preliminary results showed that regular gemcitabine administration (1000mg/m2, day 1, 8, 15 every 4 weeks) after hemihepatectomy was too toxic and induced severe leukocytopenia and/or thrombocytopenia. Formerly, the investigators planned the study to decide more safety adjuvant protocol (recommend dose: RD) for Gemcitabine or S-1 after hemihepatectomy using Continuous Reassessment Method (CRM) analysis and decided the recommend doses. Note: In the former study, the investigators decided that tolerable ratio of Dose Limiting Toxicity (DLT) would be less than 10%.

Herein, the investigators planned the study to evaluate efficacy (recurrent free survival as primary outcome, and overall-survival as secondary outcome) and safety (as secondary outcome) in our recommended protocols, and to compare the efficacy as randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. Biliary tract cancer (BTC) (>= Unio Internationalis Contra Cancrum (UICC) Stage IB), adenocarcinoma
2. R0 or R1 resection
3. no obvious recurrent lesion
4. 20 years old or more
5. Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1
6. The patient underwent no other treatment than surgery for BTC
7. Neutrophil must be over 1500/μl, Hemoglobin must be over 9.0g/dL, platelet must be over 100,000/μl, Aspartate transaminase (AST) and Alanine aminotransferase (ALT) must be less than 150 IU/L, total bilirubin must be less than 1.5 mg/dL, Creatinine must be less than 1.2 mg/dl, and Creatinine clearance must be over 60 mL/min
8. The patient can intake drugs per os.
9. From 4 to 12 weeks after the surgery
10. Written informed consent

Exclusion Criteria:

1. Existence of active double cancer
2. The patient suffered from severe drug allergy
3. Sever complications (interstitial pneumonia, heart failure, renal failure, liver failure, ileus, incontrollable diabetes mellitus, and so on)
4. Any active infections exist.
5. Pregnancy
6. Severe mental disorder
7. Others

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
1 year recurrent free survival rate | One year
  Duration: From randomization to evidenced recurrence or death. Rate: Number of patients with evidenced recurrence or death / number of total patients.
  1 year recurrent free survival rate: recurrent free survival rate at one-year from the randomization

SECONDARY OUTCOMES:
Two-year recurrent free survival rate | Two years
One-year overall survival rate | One year
Two-year overall survival rate | Two years
Completion rate of the protocol treatment | 6 months
Dose intensity of anti-tumor drugs | 6 months
Rate and grade of adverse events or adverse drug reactions | 6 months
Duration of recurrent free survival | an expected average of 2 years
Duration of overall survival | an expected average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Nagano, MD, PhD, Study Director — Osaka University Graduate School of Medicine
Locations (1):
- Osaka University, Graduate School of Medicine, Osaka, Japan